CLINICAL TRIAL: NCT00770042
Title: A Phase I, Single-Centre, Open-Label, Randomized, One-sequence Crossover, Three-Group Study to Evaluate the Effect of Ketoconazole, Ritonavir and Erythromicin on the Safety and Pharmacokinetics of Avanafil (TA-1790) in Healthy Male Subjects
Brief Title: To Evaluate The Effect Of Ketoconazole, Ritonavir and Erythromycin on the Safety and Pharmacokinetics of Avanafil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Wesley Day, VP Clinical, Vivus, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TA-011
Record Dates: First submitted 2008-10-06; First posted 2008-10-09 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-11

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Ritonavir; Ketoconazole; eryF protein, Saccharopolyspora erythraea; avanafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Ketoconazole 400 mg qd for 5 days (Days 2-6) plus a single dose of 50 mg avanafil on Days 1 and 6
  Interventions: Drug: Ketoconazole; Drug: Avanafil
- Group 2 (Experimental): Erythromycin 500mg every 12 hours for 5 days (Days 2-6) plus a single dose of 200 mg Avanafil on Days 1 and 6.
  Interventions: Drug: Erythomycin; Drug: Avanafil
- Group 3 (Experimental): Ritonavir 300 mg bid for 1 day (Day 2), 400 mg bid for 1 day (Day 3), 600 mg bid for 5 days (Day 4-8) plus a single dose of 50 mg avanafil on Days 1 and 8
  Interventions: Drug: Ritonavir; Drug: Avanafil

INTERVENTIONS:
Drug: Ritonavir — Ritonavir 300 mg bid for 1 day (Day 2), 400 mg bid for 1 day (Day 3), 600 mg bid for 5 days (Day 4-8)
  Arms: Group 3
Drug: Ketoconazole — Ketoconazole 400 mg qd for 5 days (Days 2-6)
  Arms: Group 1
Drug: Erythomycin — Erythromycin 500 mg every 12 hours for 5 days (Days 2-6)
  Arms: Group 2
Drug: Avanafil — Avanafil 50 mg on Days 1 and 8
  Arms: Group 3
Drug: Avanafil — Avanafil 50 mg on Days 1 and 6
  Arms: Group 1
Drug: Avanafil — Avanafil 200mg Days 1 and 6
  Arms: Group 2

SUMMARY:
This study is being conducted to examine the effect of three CYP3A4 inhibitors (ketoconazole, erythromycin and ritonavir) on the single dose pharmacokinetics of avanafil. Ketoconazole and ritonavir are potent inhibitors of CYP3A4 and erythromycin is a moderate CYP3A4 inhibitor. Any interaction that is observed would be predictive of other inhibitors of CYP3A4.

DETAILED DESCRIPTION:
Rationale:

Erectile dysfunction (ED) is the persistent or recurrent inability to attain and maintain penile erection sufficient to permit satisfactory sexual performance. The current first-line treatment for ED consists of oral therapy with phosphodiesterase type 5 (PDE5) inhibitors. These drugs prevents the hydrolysis of cyclic guanosine monophosphate (cGMP), resulting in increased levels of cGMP and decreased Ca+2 concentrations in the smooth muscle cells of the erectile tissues, smooth muscle relaxation and increased blood flow into the penis. The drugs are extensively metabolized in human liver microsomes, and involve the cytochrome P450, CYP2C subfamily and CYP3A4. This enzyme system is readily inhibited by many drugs. When enzymes that metabolize PDE5 inhibitors are inhibited, there may be increased plasma concentrations of the drugs and possible increases in or prolongation of therapeutic and/or adverse effects.

Avanafil is a potent and highly specific PDE5 inhibitor that is rapidly absorbed from the gastrointestinal tract and that has a relatively short half-life (0.55-1.2 hours). The formation of the main metabolites of avanafil is catalyzed by CYP3A4. It is possible that the pharmacokinetics of avanafil may be modified by drugs that block the cytochrome P450 enzyme pathways, resulting in significant changes in its pharmacokinetic (PK), efficacy and adverse event profiles. This study is being conducted to examine the effect of three CYP3A4 inhibitors (ketoconazole, erythromycin and ritonavir) on the single dose pharmacokinetics of avanafil.

Ketoconazole and ritonavir are potent inhibitors of CYP3A4 and erythromycin is a moderate CYP3A4 inhibitor. Any interaction that is observed would be predictive of other inhibitors of CYP3A4

ELIGIBILITY:
Inclusion Criteria:

1. Males, 21 to 45 years of age (inclusive).
2. A body weight of at least 50 kg and a body mass index (BMI) between 21 and 28 kg/m2, inclusive
3. Medically healthy, with clinically insignificant screening results [e.g., laboratory profiles, medical histories, ECGs, physical exam, etc., in the opinion of the investigator.
4. Subjects are able to communicate with the investigator, and to understand and comply with all requirements of study participation.
5. Voluntarily consent to participate in the study
6. The subject must agree not to donate his sperm during and within 3-months of the completion of the study.
7. All sexually active male subjects and their female partners of childbearing potential must agree to use adequate contraception methods, for the specified time.

Exclusion Criteria:

1. A history or presence of significant cardiovascular, neurological, hematological, psychiatric, hepatic, gastrointestinal, pulmonary, endocrine, immunologic or renal disease or other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs or place the subjects at increased risk as determined by the investigator.
2. Any clinically significant laboratory abnormalities as judged by the investigator.
3. Systolic blood pressure < 90 or >140 mmHg; diastolic blood pressure < 50 or > 90 mmHg at screening or at check-in on day 1 in treatment period 1.
4. Positive urine drug test and/or positive breath alcohol test.
5. Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV) at screening.
6. Any history or presence of alcoholism or drug or substance abuse.
7. Allergy to or previous adverse events with PDE5 inhibitors, ketoconazole, ritonavir and/or erythromycin or their constituents.
8. Use of any prescription or over-the-counter (OTC) medication, including herbal products.
9. Use of any drugs known to have clinical significance in inhibiting or inducing liver enzymes involved in drug metabolism
10. Blood donation or significant blood loss.
11. Any use of tobacco or nicotine products within 6 months.
12. Any history of celiac diseases, food allergies, and those on vegetarian or other diets incompatible with study objectives.
13. Any subject who received an investigational drug within 30 days .
14. Clinical judgment by the investigator that the subject should not participate in the study.

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2008-10; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of avanafil when administered with Ketoconazole, ritonavir, or erythromycin and to assess the effect of co-administration of these drugs on the pharmacokinetics of avanafil | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Shiyin Yee, PhD, Study Director — VIVUS LLC
Locations (1):
- Research Site, Lincoln, Nebraska, United States